CLINICAL TRIAL: NCT03872219
Title: The Effect of Plant and Soil-based Material on the Incidence of Atopic Sensitization
Brief Title: Biodiversity Intervention and Atopic Sensitization
Acronym: PREVALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Tampere University (Other); Pirkanmaa Hospital District (Pirkanmaan sairaanhoitopiiri) (Unknown); Business Finland (National Innovation Agency) (Unknown)
Responsible Party: Principal Investigator, Aki Sinkkonen, University Researcher, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HelsinkiUAdele2poc
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Atopy; Allergy; Allergic Rhinitis; Allergic Sensitisation
Keywords: biodiversity intervention; IgE; atopy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: The study consists of two arms, the intervention arm and the placebo arm. Children are randomized into the arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The children will receive and they are exposed daily to harmless materials that look and feel like the biodiversity intervention materials.
  Interventions: Combination Product: Nature-based materials
- intervention arm (Experimental): The children will receive and they are exposed daily to materials of high microbiological biodiversity.
  Interventions: Combination Product: Nature-based materials

INTERVENTIONS:
Combination Product: Nature-based materials — In the intervention arm, theycontain inactive and slowly-growing environmental bacteria and other microbiota. In the placebo arm, they do not contain the microbiota.

SUMMARY:
Children will receive biodiversity intervention or placebo. The proof of concept trial is double blind. Intervention will start at the age of 2 months and last 10 months. Children will be randomized to arms. IgE sensitization is the primary outcome.

DETAILED DESCRIPTION:
Newborns will start to be exposed to biodiversity intervention or placebo at the age of two months. The proof of concept trial will be double blind. Intervention will start at the age of 2 months and it will end when children become 12 months old. Children will be randomized to the two arms. IgE sensitization is the primary outcome at the age of two and three years.

ELIGIBILITY:
Inclusion Criteria:

* both parents have atopy
* newborn

Exclusion Criteria:

* severe disease, particularly immune system deficiency or down syndrome or cancer
* medication affecting immune system
* birth before week 35 in pregnancy
* being a twin
* only one of the parents have atopy
* none of the parents have atopy
* children have passed the age of two months
* immune system disorder such as rheumatoid disease, colitis ulcerosa, Crohn disease, diabetes or genetic risk to type 1 diabetes
* no participation in national vaccination programme

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
IgE sensitization | 2-3 years
  IgE sentitization is expected to be lower in the intervention arm than in the placebo arm.

SECONDARY OUTCOMES:
Allergic symptoms | 2-3 years
  All possible allergic symptomes, including atopy, will be estimated

OTHER OUTCOMES:
IL-10: IL-17 ratio | 2-3 years
TGF-beta level | 2-3 years
IL-10 levels | 2-3 years

IPD SHARING:
Plan to Share IPD: No
We will share it according to Finnish legislation and ethical committee permission. The permission restrict sharing tightly.